CLINICAL TRIAL: NCT01624168
Title: Effects of Tai Chi Chuan on Psychobiological Indicators of Anxiety and Sleep Quality in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Principal Investigator, Karen Caldwell, Professor, Appalachian State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBT Feasibility
Record Dates: First submitted 2012-06-15; First posted 2012-06-20 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Anxiety
Keywords: anxiety; sleep quality; tai chi chuan; young adults
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anxiety Management Education (Placebo Comparator)
  Interventions: Behavioral: Anxiety Management Education
- 10 week tai chi intervention (Experimental): 10 week course in Evidence Based Tai Chi meeting 2 times per week
  Interventions: Behavioral: 10 week tai chi intervention
- Enhanced tai chi instruction (Experimental): 10 weeks of instruction in Evidence Based Tai Chi meeting 2 times per week plus DVD for home practice
  Interventions: Behavioral: Enhanced tai chi instruction

INTERVENTIONS:
Behavioral: Anxiety Management Education — written materials on management of anxiety for self-study
  Arms: Anxiety Management Education
Behavioral: 10 week tai chi intervention — 10 weeks of instruction in Evidence Based Tai Chi meeting 2 times per week
  Arms: 10 week tai chi intervention
Behavioral: Enhanced tai chi instruction — 10 weeks of instruction in Evidence Based Tai Chi meeting 2 times per week plus DVD for home practice
  Arms: Enhanced tai chi instruction

SUMMARY:
The purpose of this study is to determine the feasibility of a 10-week tai chi chuan intervention as a treatment for anxiety and sleep quality in young adults.

ELIGIBILITY:
Inclusion Criteria:

* mild to severe symptoms of anxiety
* interest in participating in an exercise intervention
* willingness to accept randomization
* provides informed consent
* low or moderate risk for acute cardiovascular event

Exclusion Criteria:

* currently receiving psychotherapy or medication for psychological problems
* current suicide or homicide risk
* current or history of psychosis
* current alcohol or substance dependence
* high risk for an acute cardiovascular event
* current use of prescription drugs with potential to influence the parasympathetic or sympathetic nervous system
* current or previous extensive involvement in mind-body exercise
* symptoms of severe depression

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L. Caldwell, PhD, Principal Investigator — Appalachian State University
Locations (1):
- Appalachian State University, Boone, North Carolina, United States

REFERENCES:
- [Background] Caldwell K, Harrison M, Adams M, Quin RH, Greeson J. Developing mindfulness in college students through movement-based courses: effects on self-regulatory self-efficacy, mood, stress, and sleep quality. J Am Coll Health. 2010 Mar-Apr;58(5):433-42. doi: 10.1080/07448480903540481. PMID 20304755
- [Background] Caldwell K, Harrison M, Adams M, Triplett NT. Effect of Pilates and taiji quan training on self-efficacy, sleep quality, mood, and physical performance of college students. J Bodyw Mov Ther. 2009 Apr;13(2):155-63. doi: 10.1016/j.jbmt.2007.12.001. Epub 2008 Feb 20. PMID 19329051
- [Background] Caldwell K, Emery L, Harrison M, Greeson J. Changes in mindfulness, well-being, and sleep quality in college students through taijiquan courses: a cohort control study. J Altern Complement Med. 2011 Oct;17(10):931-8. doi: 10.1089/acm.2010.0645. Epub 2011 Oct 14. PMID 21999153

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction
Started | 19 | 28 | 28
Completed | 15 | 16 | 22
Not Completed | 4 | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction | Total
Number analyzed (Participants) | 19 | 28 | 28 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.42 (5.47) | 21.21 (3.04) | 20.18 (1.16) | 21.13 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 19 | 51
  Male | 5 | 10 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Retention of Randomized Subjects During Intervention
Description: Retained subjects are those who are willing to return for complete assessments
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction
Number analyzed (Participants) | 19 | 28 | 28
participants
  Retained | 17 | 22 | 25
  Not retained | 2 | 6 | 3

2. Primary Outcome: Retention of Randomized Subjects for Follow-up
Description: Subjects retained for follow-up are those willing to respond to follow-up assessments
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction
Number analyzed (Participants) | 19 | 28 | 28
participants
  Retained for follow-up | 15 | 16 | 22
  Lost to follow-up | 4 | 12 | 6

3. Primary Outcome: Adherence to Out-of-class Practice
Description: Subjects are considered adherent to out-of-class practice if he/she practices outside of class twenty times during the 10 week intervention
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction
Number analyzed (Participants) | 19 | 28 | 28
participants
  Adherent to out-of-class practice | NA — Individuals in the Anxiety Management Education group did not participate in tai chi classes or home practice. | 13 | 20
  Not adherent to out-of-class practice | NA — Individuals in the Anxiety Management Education group did not participate in tai chi classes or home practice. | 15 | 8

4. Primary Outcome: Adherence to Practice After the Intervention
Description: Subjects are considered adherent to practice after the intervention if they practice an average of 2 times per week.
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction
Number analyzed (Participants) | 19 | 28 | 28
participants
  Adherent to practice after the intervention | NA — Individuals in the Anxiety Management Education group did not participate in tai chi classes or home practice. | 4 | 13
  Not adherent to practice after the intervention | NA — Individuals in the Anxiety Management Education group did not participate in tai chi classes or home practice. | 24 | 15

5. Secondary Outcome: Change From Baseline in State Anxiety Scores
Description: Anxiety was measured by the State Trait Anxiety Inventory - State Scale. Lower scores on this scale reflect better outcomes. Scores can range from 20 to 80.
Time Frame: change from baseline to 4 weeks, 10 weeks, 2 month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction
Number analyzed (Participants) | 17 | 22 | 25
units on a scale
  Change from Baseline to 4 weeks | -1.93 (2.06) | -2.70 (1.79) | -3.17 (1.68)
  Change from Baseline to 10 weeks | -1.43 (2.09) | -4.36 (1.89) | -3.04 (1.73)
  Change from Baseline to 2 Month Follow-up | -1.90 (2.15) | -5.08 (2.03) | -3.58 (1.78)

6. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index Scores
Description: Sleep quality was measured by the Pittsburgh Sleep Quality Index Total Score. Lower scores on this scale reflect better outcomes. Scores can range from 0 to 21.
Time Frame: baseline, 4 weeks, 10 weeks, 2 month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction
Number analyzed (Participants) | 17 | 22 | 25
units on a scale
  Change from Baseline to 4 weeks | -1.06 (.45) | -1.40 (.39) | -1.32 (.36)
  Change from Baseline to 10 weeks | -1.71 (.46) | -2.98 (.41) | -2.03 (.38)
  Change from Baseline to 2 month follow-up | -1.82 (.47) | -3.60 (.45) | -3.05 (.38)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were asked to complete weekly reports of mood using the Generalized Anxiety Disorder-7 scale and the Patient Health Questionnaire - 2. Participants also were asked about adverse events at 4-week and 10-week laboratory visits.
Arm/Group | Anxiety Management Education | 10 Week Tai Chi Intervention | Enhanced Tai Chi Instruction
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/28 | 1/28
Other Adverse Events (participants affected / at risk) | 9/19 | 9/28 | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anxiety Management Education (N=19) | 10 Week Tai Chi Intervention (N=28) | Enhanced Tai Chi Instruction (N=28)
overdose suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Fell on ice, broke ankle (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anxiety Management Education (N=19) | 10 Week Tai Chi Intervention (N=28) | Enhanced Tai Chi Instruction (N=28)
Anger (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 1 | 3
Anxiety with Depression (Psychiatric disorders) | 2 | 1 | 1
Cold (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Family Stress (Social circumstances) | 2 | 0 | 1
Feeling Blue (Psychiatric disorders) | 0 | 2 | 4
Feeling sick (General disorders) | 0 | 2 | 3
Knee pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Poor sleep (Nervous system disorders) | 1 | 0 | 1
Stress (Psychiatric disorders) | 1 | 1 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1
Worry (Psychiatric disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
None of the reported Serious Adverse Events or Adverse Events were determined to be a result of participation in the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No